CLINICAL TRIAL: NCT04533295
Title: The Effect of Acupuncture on IVF Pregnancy Outcomes for Women With Recurrent Implantation Failure: a Multi-center Randomized Controlled Clinical Trial
Brief Title: The Effect of Acupuncture on IVF Pregnancy Outcomes for Women With RIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Cui Hong Zheng, associate professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019CR110
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Repeated Implantation Failure
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture and IVF (Experimental): Acupuncture and IVF
  Interventions: Device: acupuncture and IVF
- Sham acupuncture and IVF (Sham Comparator): Sham acupuncture and IVF
  Interventions: Device: sham acupuncture and IVF

INTERVENTIONS:
Device: acupuncture and IVF — Acupuncture was performed three times a week for 30 minutes each time, starting from the 5th day of menstruation and ending within 24 hours after embryo transfer.
  Arms: Acupuncture and IVF
Device: sham acupuncture and IVF — Sham acupuncture was performed three times a week for 30 minutes each time, starting from the 5th day of menstruation and ending within 24 hours after embryo transfer.
  Arms: Sham acupuncture and IVF

SUMMARY:
The randomized, placebo-controlled multicenter trial is conducted in five centers in China. After screening and obtaining the signed informed consent , the participants are randomly divided into two groups: acupuncture +IVF group and sham acupuncture +IVF group.

ELIGIBILITY:
Inclusion Criteria:

1. Married women aged 25-40;
2. Repeated implantation failure for unknown reasons (after 3 or more consecutive cycles of embryo transfer, or cumulative transfer of ≥6 high-quality cleavage embryos or 4 high-quality blastocysts without clinical pregnancy);
3. Transplantable Day 3 high-quality frozen embryos or frozen blastocysts (≥3BB);
4. Estrogen and progesterone replacement therapy (HRT), endometrial thickness ≥7mm on the day of endometrial transformation.

Exclusion Criteria:

Patients who met any of the following conditions were not included.

1. Those who prepare for PGD;
2. Recipients of egg donors;
3. Chromosomal abnormalities in both or one of the couples (excluding chromosome polymorphism);
4. patients with implantation failure due to known embryonic factors;
5. Uterine lesions that may affect implantation (including uterine malformation, uterine tuberculosis, history of intrauterine adhesions, submucosal fibroids, adenomyosis, >4cm intramural fibroids)
6. Repeated spontaneous abortion (2 or more fetal loss before 28 weeks of gestation);
7. Patients with other endocrine diseases, such as thyroid disease, hyperprolactinemia, insulin resistance, diabetes, adrenal disease, etc., and poor control of hormone levels in the last 3 months;
8. Clearly diagnosed autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid syndrome, etc.;
9. Hydrosalpinx untreated;
10. BMI less than 18 and higher than 25kg/m2;
11. People with previous history of needle sickness;
12. Those who had previously participated in this study or had received acupuncture treatment in the past 3 months.
13. Any situation that researchers consider inappropriate for participating in this study.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 514 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CPR | 1 month after ET
  Clinical pregnancy rate

SECONDARY OUTCOMES:
OPR | 3 month after ET
  ongoing pregnancy rate
LBR | 10 month after ET
  Live birth rate
Biochemical indexes | one year
  Biochemical indexes
Questionnaire score | one year
  Questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Minming Zhang, professor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital,Tongji medical college,HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No